CLINICAL TRIAL: NCT04648826
Title: Phase I/II Evaluation of Aerosolized Azacytidine as Epigenetic Priming for Bintrafusp Alfa-Mediated Immune Checkpoint Blockade in Patients With Unresectable Pulmonary Metastases From Sarcomas, Germ Cell Tumors, or Epithelial Malignancies
Brief Title: Aerosolized Azacytidine as Epigenetic Priming for Bintrafusp Alfa-Mediated Immune Checkpoint Blockade in Patients With Unresectable Pulmonary Metastases From Sarcomas, Germ Cell Tumors, or Epithelial Malignancies
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to notification from EMD Serono, for Bintrafusp alfa (M7824) regarding an observed increase in the frequently of early progression and death.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 210004; 21-C-0004
Record Dates: First submitted 2020-12-01; First posted 2020-12-02 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Sarcomas; Melanomas; Germ Cell Tumors; Epithelial Malignancies (Excluding Lung and Renal Cell Carcinomas); Pulmonary Metastases
Keywords: M7824; AZA; unresectable pulmonary metastases; inhalational epigenetic priming regimen; aerosol drug delivery
MeSH Terms: conditions — Sarcoma; Melanoma; Neoplasms, Germ Cell and Embryonal; Carcinoma, Renal Cell | interventions — bintrafusp alfa protein, human; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/ Phase I Dose Escalation (Experimental): Azacytidine (aerosolized) at escalating doses (given on 3 consecutive days in the first week of every 3-week cycle) with a flat dose of Bintrafusp alfa 2400 mg (given on day 13 [+/- 3 days] of every 3-week cycle starting with Cycle 2)
  Interventions: Device: AeroEclipse II Breath Actuated Nebulizer; Drug: Bintrafusp alfa; Drug: Azacytidine
- 2/ Phase II Dose Expansion (Experimental): Azacytidine (aerosolized) at the RP2D established in Phase I (given on 3 consecutive days in the first week of every 3-week cycle) with a flat dose of Bintrafusp alfa 2400 mg (given on day 13 [+/- 3 days] of every 3-week cycle)
  Interventions: Device: AeroEclipse II Breath Actuated Nebulizer; Drug: Bintrafusp alfa; Drug: Azacytidine

INTERVENTIONS:
Device: AeroEclipse II Breath Actuated Nebulizer — Patients will receive AZA via commercial device, AeroEclipse II Breath Actuated Nebulizer.
Drug: Bintrafusp alfa — Bintrafusp alfa will be administered on Day 13 (+/- 3 days) of every 3-week cycle (i.e., Q3W [once every 3 weeks]) at a fixed intravenous dose of 2400 mg; Bintrafusp alfa does not start until cycle 2 of the phase I portion.
Drug: Azacytidine — Patients will receive azacytidine (aersolized; via commercial AeroEclipse II Breath Actuated Nebulizer device) on 3 consecutive days in the first week of every 3-week cycle. Phase I: Azacytidine will be given at escalating doses. Phase II: Azacytidine will be given at the RP2D established in Phase I.

SUMMARY:
Background:

About one-third to one-half of all people dying of extrathoracic malignant diseases have cancer that has spread to the lungs. Surgery may help some people. But most people with pulmonary metastases do not survive long. Researchers want to see if a combination of drugs can help.

Objective:

To find a safe dose of Azacytidine, when taken as a fine mist that is inhaled (aerosolized Azacytidine), together with Bintrafusp Alfa to treat cancers that have spread to the lungs.

Eligibility:

Adults ages 18 and older who have cancer that has spread to the lungs, cannot be cured with surgery, and has not responded to standard treatments.

Design:

Participants will get Azacytidine by breathing treatments once a day for 3 days each week, for 3 weeks. The 3-week period is 1 cycle. Each course of treatment is 3 cycles.

Once per cycle, participants will get Bintrafusp Alfa via IV. An IV is a small tube that is put into an arm vein.

Participants will keep a diary of any side effects.

Participants can take the study drugs for as long as they can continue treatment.

Participants will have medical histories and physical exams. They will give blood, urine, and lung lining fluid samples. Tumor samples will be taken via bronchoscopy. They will have lung function tests.

Participants will have an imaging scan that shows how spray particles move in their airway when they inhale. They will have tumor imaging scans of the chest and brain.

Participants will have a follow-up visit 30 days after they stop treatment....

DETAILED DESCRIPTION:
Background:

While malignancies of diverse histologies express a variety of cancer-testis antigens (CTAs), immune responses to these proteins appear uncommon in cancer patients due to low-level, heterogeneous antigen expression, as well as local and systemic immunosuppression.

CTAs such as NY-ESO-1 and MAGE-A3 can be up-regulated in tumor cells of various histologies, but not in normal cells, by DNA demethylating agents such as decitabine (DAC) and azacytidine (AZA). Up-regulation of these CTAs facilitates CTL-mediated lysis of tumor cells.

Clinical trials have demonstrated impressive regressions of tumors expressing NY-ESO-1 following adoptive immunotherapy targeting this CTA.

In addition to shared CTAs, unique neoantigens are major targets for immune eradication of cancer cells.

DNA demethylating agents not only up-regulate cancer-testis (CT) genes but also induce expression of endogenous retroviruses (ERV) which further augments immunogenicity of cancer cells.

Additionally, DNA demethylating agents enhance antigen processing and presentation by cancer cells, and inhibit activity of myeloid derived suppressor cells (MDSC), thereby increasing the efficacy of immune checkpoint inhibitors in murine tumor models.

Despite these provocative preclinical results, epigenetic priming for immune checkpoint blockade has yet to be translated to humans due to systemic toxicities and pharmacokinetic/pharmacodynamic limitations that prevent optimal dosing of DNA demethylating agents.

One potential strategy to enhance delivery of DNA demethylating agents to pulmonary malignancies while minimizing systemic toxicities is to administer these drugs by inhalation techniques.

Preclinical studies have demonstrated that aerosolized AZA mediates epigenetic activation of gene expression in orthotopic lung cancers, and significantly prolongs survival of mice bearing these tumors without systemic toxicities.

Conceivably, inhaled AZA may help to prime pulmonary malignancies for immune checkpoint blockade.

In this study, the optimal dose of inhaled AZA will be established in patients with unresectable pulmonary metastases who are receiving the dual immune checkpoint inhibitor-TGF-Beta trap, Bintrafusp alfa (M7824).

This trial is intended to establish the rationale for further evaluation of inhalational epigenetic priming regimens in combination with immune checkpoint inhibitors or adoptive cell transfer regimens in patients with locally advanced pulmonary malignancies.

Objectives:

Phase I component: To determine pharmacokinetics, toxicities, maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of aerosolized AZA in patients receiving Bintrafusp alfa for unresectable pulmonary metastases

Phase II component: To determine frequency of intrathoracic clinical responses in these patients following administration of aerosolized AZA at the RP2D and Bintrafusp alfa.

Both components: To determine safety of aerosolized AZA and Bintrafusp alfa in patients with unresectable pulmonary metastases.

Eligibility Criteria:

Patients with histologically or cytologically proven, unresectable pulmonary metastases from sarcomas, melanomas, germ cell tumors, or epithelial malignancies (except lung or kidney cancers) who have received first line standard of care treatment for their metastatic disease.

Measurable disease by RECIST

Patients are eligible irrespective of intratumoral PD-L1 expression.

Patients with prior treatment with an immune checkpoint inhibitor and DNA demethylating agents may be eligible for study provided they did not experience serious immune adverse events that required discontinuation of the drug, and more than three weeks have elapsed since treatment

Patients greater than or equal to 18 years; ECOG performance status of 0-1 without evidence of unstable or decompensated myocardial disease; adequate pulmonary reserve evidenced by FEV1 greater than or equal to 60% predicted, FEV1/FVC ratio greater than or equal to 60%, and adjusted DLCO greater than or equal to 60% predicted; pCO2 less than or equal to 45 mm Hg and pO2 greater than or equal to 60 mm Hg on room air ABG

Adequate renal, hepatic and hematopoietic function

Design:

Subjects will receive aerosolized AZA on three consecutive days (i.e.; Days 1, 2, and 3, or Days 3, 4, 5) of a 21-day cycle. Three cycles constitute one course of treatment.

Bintrafusp alfa will be administered at a fixed dose of 2400 mg. During Phase I, Bintrafusp alfa will be administered on Day 13 (i.e., once every 3 weeks, one week after AZA) of each cycle starting from Cycle 2 of Course 1 (i.e., no Bintrafusp alfa in the first cycle of Course 1). During Phase II, Bintrafusp alfa will be administered the day after the last AZA treatment, during Week 1 of each treatment cycle.

The dose of AZA will be escalated during Phase I using a 3+3 design with no intrapatient dose escalation.

The dose of AZA will be sequentially increased to maximize intra-tumoral DNMT1 depletion while avoiding Grade 3 or greater pulmonary or systemic toxicities attributable to this agent during the first cycle of therapy.

Treatment evaluation will be three weeks +/- one week following completion of each course of therapy.

Once the RP2D of aerosolized AZA has been defined, that dose level will be expanded to a total of 9 patients to determine response rates at the RP2D using a Simon two stage design for Phase II trials.

Approximately 42 patients will be accrued to this trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Histologically or cytologically confirmed, unresectable pulmonary metastases from sarcomas, melanomas, germ cell tumors, or epithelial malignancies excluding lung and renal cell carcinomas.
  2. Patients with extrathoracic disease may be eligible provided there are 5 or fewer low volume non-thoracic sites (less than or equal to 3 cm/nodule) that are not life-threatening and are potentially treatable with metastasis-directed therapy whether they are symptomatic or not.
  3. Patients with bone metastases (less than 5 sites) are potentially eligible for study.
  4. Patients must have received first line standard of care systemic treatment for their malignancies.
  5. Patients with tumors with potentially actionable mutations are eligible for study if their metastases are refractory to approved first-line targeted agents.
  6. Patient's PD-L1 expression in cancer cells may be positive or negative as quantitated by immunohistochemistry techniques.
  7. Patients must have measurable disease per RECIST 1.1.
  8. Patient's pulmonary disease can be safely accessed via bronchoscopic, thoracoscopic or transthoracic percutaneous biopsy, and patient must be willing to undergo biopsy as well as bronchoscopy before and after treatment.
  9. Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of aerosolized AZA in patients < 18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.
  10. ECOG performance status of less than or equal to 1
  11. Patients must be without evidence of unstable or decompensated myocardial disease, and have adequate pulmonary reserve evidenced by FEV1 and adjusted DLCO greater than or equal to 60% predicted and FEV1/FVC ratio greater than or equal to 60%; pCO2 less than or equal to 45 and pO2 greater than ir equal to 60 on room air.
  12. Normal organ and marrow function as defined below:

      * leukocytes greater than or equal to 3,000/mcL
      * absolute neutrophil count greater than or equal to 1,500/mcL (without transfusion or cytokine support)
      * absolute lymphocyte count > 800/mcL
      * platelets greater than or equal to 100,000/mcL
      * Hgb greater than or equal to 9 g/ dL
      * PT no more than 2 seconds above the ULN
      * total bilirubin < 1.5 X institutional upper limit of normal

      OR
      * direct bilirubin less than or equal to ULN for patients with total bilirubin > 1.5 ULN
      * serum albumin greater than or equal to 2.0 mg/dL
      * AST(SGOT)/ALT(SGPT) less than or equal to 1.5 X institutional ULN
      * ALP less than or equal to 2.5 X institutional ULN
      * creatinine less than or equal to 1.6 mg/mL

      OR

      --creatinine clearance (eGFR) greater than or equal to 30 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal

      at the time AZA and M7824 treatment commences.
  13. Patients with history of brain metastases except those with meningeal carcinomatosis or leptomeningeal disease may be eligible for treatment a minimum of 2 weeks following completion of gamma knife or whole brain radiotherapy, or 4 weeks following surgical resection of brain metastasis; provided post-treatment MR scan reveals no evidence of active disease, and no ongoing need for systemic steroids.
  14. The effects of AZA and Bintrafusp alfa on the developing human fetus are unknown. For this reason and because the agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 125 days following the last dose of Bintrafusp alfa for males, and 65 days following the last dose of Bintrafusp alfa for females.
  15. Ability of subject to understand and the willingness to sign a written informed consent document.
  16. Ability of subject and the willingness to co-enroll and sign a written informed consent document for 06C0014 "Prospective Evaluation of Genetic and Epigenetic Alterations in Patients with Thoracic Malignancies".

EXCLUSION CRITERIA:

1. Patients with cancers harboring mutations targetable with approved agents who have not progressed on targeted therapy.
2. Patients with primary lung cancers are excluded from study due to potential exacerbation of pulmonary toxicities from investigational therapy due to evolution or treatment of their malignancies.
3. Patients with renal cancers are excluded from study due to potential bleeding from these highly vascular metastases.
4. Active smokers
5. Patients either receiving systemic steroids other than physiologic replacement doses, or inhaled corticosteroids.
6. Previous treatment with targeted therapy, immune checkpoint inhibitor, DNA demethylating agent, systemic chemotherapy, or radiation therapy to an index lesion within three weeks prior to starting protocol therapy. Patients with prior treatment with immune checkpoint inhibitors, and DNA demethylating agents may be eligible for study provided more than three weeks have elapsed since treatment and they did not experience serious immune adverse events that required discontinuation of the immune checkpoint

   inhibitor.
7. History of allergic reactions attributed to compounds of chemical or biologic composition similar to Bintrafusp alfa and AZA.
8. Clinically significant cardiovascular / cerebrovascular disease as follows: cerebral vascular accident / stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class greater than or equal to II), serious cardiac arrhythmia, clinically significant bleeding or clinically significant pulmonary embolism.
9. History of pneumonitis (idiopathic or drug induced) unless cleared by pulmonary consultants.
10. Receipt of any organ transplantation, including allogeneic stem-cell transplantation, except for transplants that do not require immunosuppression (e.g., corneal transplant, hair transplant).
11. Active Hepatitis A, Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
12. Human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness due to unknown effects of AZA on systemic immunity.
13. Other active infection requiring systemic therapy, including COVID-19 (testing will be required as part of screening).
14. Pregnant women are excluded from this study because AZA and Bintrafusp alfa may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Bintrafusp alfa and AZA, breastfeeding should be discontinued if the mother is treated with Bintrafusp alfa and AZA.
15. Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
16. Recent major bleeding events considered by the Investigator as high risk for investigational drug treatment.
17. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent with the exceptions:

    * Diabetes type I, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment;
    * Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses less than or equal to 10 mg of prednisone or equivalent per day;
    * Administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or intra-articular).
18. Patients receiving another investigational agent.
19. An additional malignancy that is progressing or requires active treatment.
20. Administration of live vaccines with 30 days prior to enrollment. Administration of inactivated vaccines (e.g., inactivated influenza vaccines) is permitted during the study.
21. Subjects unwilling to accept blood products as medically indicated.
22. Emotional, psychiatric or substance abuse disorders that would interfere with cooperation with the requirements and safety of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Phase I: Determine pharmacokinetics, toxicities, maximum tolerated dose and recommended Phase 2 dose (RP2D) of aerosolized AZA in patients receiving IV Bintrafusp alfa for unresectable pulmonary metastases | baseline, first treatment, end of each course
  DLTs at each Phase I dose level will be reported. Pharmacokinetic analysis will be conducted using non-compartmental methods. All patients will be evaluable for toxicity from the time of their first treatment with AZA/ Bintrafusp alfa. Dose limiting toxicities will be assessed during the first 3 cycles of AZA/ Bintrafusp alfa therapy. Patients who have measurable disease present at baseline, have received at least 9 weeks of AZA/Bintrafusp alfa therapy (three cycles), and have had their disease re-evaluated will be considered evaluable for response.
Phase II: Determine frequency of intrathoracic objective clinical response in patients with unresectable pulmonary metastases following administration of aerosolized AZA at the RP2D and IV Bintrafusp alfa | baseline, end of each course
  Patients who have measurable disease present at baseline, have received at least 9 weeks of AZA/Bintrafusp alfa therapy (three cycles), and have had their disease re-evaluated will be considered evaluable for response provided.

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2021-C-0004.html